CLINICAL TRIAL: NCT02722083
Title: A Single-blind, Randomized, Placebo Controlled, Crossover Pilot Study to Evaluate the Onset of Action of an Antihistamine in Subjects Following Allergen Exposure in an Allergen Chamber
Brief Title: Exploratory Study for Allergy Relief Onset
Status: Terminated | Phase: Phase 2 | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: 18573
Record Dates: First submitted 2016-03-23; First posted 2016-03-29 (Estimated); Last update posted 2018-12-12 (Actual); Status verified 2018-12

CONDITIONS: Rhinitis, Allergic
MeSH Terms: conditions — Rhinitis, Allergic | interventions — Chlorpheniramine

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- BAY X002134 (Experimental): Subjects will be given BAY X002134
  Interventions: Drug: Chlorpheniramine maleate (BAY X002134)
- Placebo (Placebo Comparator): Subjects will be given a placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Chlorpheniramine maleate (BAY X002134) — 4 mg tablet, single dose, orally
  Arms: BAY X002134
Drug: Placebo — placebo tablet, single dose, orally
  Arms: Placebo

SUMMARY:
The purpose of the study is to explore the onset of effect of an antihistamine in a controlled environment.

ELIGIBILITY:
Inclusion Criteria:

* Ambulatory healthy male and female subjects between 18 to 65 years of age inclusive;
* Self-reported to have seasonal allergic rhinitis for at least 2 years prior
* Documented positive skin prick test response to common ragweed (ambrosia artemisiifolia) pollen; prick with wheal > 4mm larger than the diluent within the previous 12 months
* Total Symptom Score (TSS) ≥ 40 mm at the 90 or 120 minute time point during one of the Priming Visits and at 90 or 120 minute time points during ragweed challenge Symptom Induction Phase of each Treatment Visit;
* Body Mass Index (BMI) in the range of 18 to 30 kg/m2
* Female subjects of childbearing potential must be using a medically acceptable form of birth control for at least 1 month prior to screening (3 months on oral contraceptives), e.g., oral or patch contraceptives, intrauterine device, injectable contraceptive (e.g. Depo-Provera®), or a double barrier and have a negative pregnancy test at Screening and prior to IMP administration on Day 1 and Day 7 ± 1 day. Female subjects of non-childbearing potential must be amenorrheic for at least two years or had a hysterectomy and/or bilateral oophorectomy

Exclusion Criteria:

* Evidence or self-reported history of significant medical condition which, in the judgment of the investigator, is a contraindication to the use of chlorpheniramine, or might interfere with the trial. These may include thyroid disease (e.g., hyperthyroidism, hypothyroidism), uncontrolled diabetes mellitus, coronary heart disease, ischemic heart disease , symptomatic prostatic hypertrophy, bladder neck obstruction, hepatic insufficiency, narrow-angle glaucoma, pyloroduodenal obstruction, or stenosing peptic ulcer;
* Known allergy to chlorpheniramine, dexchlorpheniramine, or any of its inactive ingredients
* Self-reported non-responders (lack of therapeutic effect) to antihistamines
* Administration of epinephrine is contra-indicated;
* Current use of oral steroids, including prednisone and prednisolone;
* Females who are pregnant or lactating
* A history of anaphylaxis to ragweed allergen
* Subjects with a history of asthma, lower respiratory tract disease, emphysema or chronic bronchitis; At the discretion of the investigator, subjects with self-reported mild intermittent asthma or exercise induced asthma may be included.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2016-05-07 (Actual); Primary Completion 2016-05-27 (Actual); Study Completion 2016-07-13 (Actual)

PRIMARY OUTCOMES:
The time to the meaningful relief, as defined by at least 15% of reduction from baseline in Total Symptom Score (TSS) | 4 hours

SECONDARY OUTCOMES:
Number of patients with adverse events as a measure of safety | 3 month

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (1):
- Germantown, Tennessee, United States